CLINICAL TRIAL: NCT05065697
Title: Brain Lesions After Transcatheter Aortic Valve Replacement
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Collaborators: St Thomas' Hospital, London (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mao Chen, Director of Department of Cardiology, West China Hospital
Other Study IDs: 2021V1
Record Dates: First submitted 2021-09-08; First posted 2021-10-04 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Aortic Valve Stenosis; Brain Diseases
Keywords: TAVR; Magnetic resonance imaging; Ischemic infarct; Microbleeds
MeSH Terms: conditions — Aortic Valve Stenosis; Brain Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TAVR arm: Symptomatic severe aortic stenosis undergoing transfemoral TAVR of any devices
  Interventions: Other: Brain MRI
- SAVR arm: Symptomatic severe aortic stenosis undergoing isolated bioprosthetic surgical aortic valve replacement
  Interventions: Other: Brain MRI

INTERVENTIONS:
Other: Brain MRI — Brain MRI will be scheduled within three days before the procedure and within seven days after the procedure, as well as at 1-year follow-up. MRI will be preferably performed using a 3.0-Tesla system unless patients are pacemaker-dependent after the procedure. In such case, a 1.5-Tesla system will be used. The MRI protocol consists of standardized conventional diffusion-weighted MRI (DW-MRI), T2-FLAIR (fluid-attenuated recovery inversion) and SWI (susceptibility-weighted imaging) parameters.
  Other Names: Neurological and cognitive assessments as recommended by NeuroARC

SUMMARY:
The Brain lEsions after TrAnscatheter aorTic ValvE Replacement (BETTER) registry is a prospective, observational, multi-center registry aiming to assess the presence of new brain microbleeds assessed on susceptibility-weighted imaging at 3 enrolling sites, in China (West China Hospital, Sichuan University), UK (St Thomas' Hospital) and Denmark (Rigshospitalet, University of Copenhagen). The main study arm is planned to include 100 patients with symptomatic severe aortic stenosis undergoing transfemoral TAVR of any devices and 50 isolated bioprosthetic SAVR patients treated during the enrollment period as a control arm.

DETAILED DESCRIPTION:
"Silent" stroke post-TAVR presents as asymptomatic brain ischemic lesions detected on diffusion-weighted magnetic resonance imaging (DW-MRI), with an incidence ranging from 60% to 100% in different studies. On the contrary, hemorrhagic lesions are not systematically studied given the poor visualization of small hemorrhage (i.e. microbleeds) on traditional T1, T2 or DW-MRI sequences. We have previously identified an incidence of new brain microbleeds early after TAVR of 100% with the routine use of susceptibility-weighted imaging (SWI). We hypothesize that new brain microbleeds are prevalent in patients with aortic stenosis after either TAVR or SAVR. The key objective of this registry is to evaluate the incidence, distribution and clinical impact of new brain microbleeds after transfemoral TAVR in patients with symptomatic severe aortic stenosis, in comparison with SAVR.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic severe aortic stenosis (>60 years old) being scheduled for either transfemoral TAVR or isolated SAVR

Exclusion Criteria:

* Patients who have been diagnosed with brain cancer, brain haemorrhage, brain abscess, aneurysm, cerebral palsy, encephalitis, nervous system infection, head or neurological injury, or trauma, stroke
* Contraindications for a magnetic resonance imaging (MRI) scan (i.e. metallic implants, claustrophobia, MR-incompatible pacemakers or prosthetic heart valves)
* Unremovable dental prostheses that are deemed to affect MRI quality
* Severe coronary artery disease that is unrevascularized
* Prior stroke within the last 12 months
* Expected non-compliance concerning follow-up examinations
* Have participated in other clinical trials

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic severe aortic stenosis (>60 years old) being scheduled for either transfemoral TAVR or isolated SAVR at enrolling sites will be invited to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of new brain microbleeds detected on MRI | Post-procedurally (up to 7 days) and 6 months
  Microbleeds (including the number and size) on SWI after TAVR or SAVR during the index hospitalization and their evolution at the follow-up
The incidence of new brain embolisms detected on MRI | Post-procedurally (up to 7 days) and 6 months
  Ischemic infarcts (including the number and size) on DW-MRI after TAVR or SAVR during the index hospitalization and their evolution at the follow-up

SECONDARY OUTCOMES:
Changes in the neurological and cognitive status of the patients (see description for specific assessments) | Post-procedurally (up to 7 days), 6 months and 1 year
  NIH Stroke Scale (NIHSS) and Montreal Cognitive Assessment (MoCA, cognitive impairment = score <23/30) for overall cognitive status, and tests for five individual cognitive domains (Attention: Digit Symbol-Coding test [DSST]; Memory: Hopkins Verbal Learning Test-Revised [HVLT-R], Brief Visual Memory Test-Revised [BVMT-R]; Executive Function: Stroop Color-Word Association Test [SCWT], Category and Verbal Fluency [both semantic and phonemic]; Visuospatial Function: BVMT-R). The change of score in each assessment will be calculated.

OTHER OUTCOMES:
Perfusion changes on transcranial doppler during TAVR or SAVR (if obtained) | Intra-procedurally
  Baseline perfusion will be obtained before femoral puncture in TAVR and the start of cardiopulmonary bypass in SAVR, until completion of eventual postimplantation maneuvers in TAVR and the stop of cardiopulmonary bypass in SAVR